CLINICAL TRIAL: NCT03956862
Title: A Phase 2a, Randomized, Double-Blind, Placebo-Controlled, Multi-Center Study to Evaluate the Effect of GB001 in Patients With Chronic Rhinosinusitis With or Without Nasal Polyps
Brief Title: GB001 in Adult Participants With Chronic Rhinosinusitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GB001, Inc, a wholly owned subsidiary of Gossamer Bio, Inc. (Industry)
Responsible Party: Sponsor
Organization: Gossamer Bio Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GB001-2101; 2019-001682-33 (EudraCT Number)
Record Dates: First submitted 2019-05-17; First posted 2019-05-21 (Actual); Results first posted 2021-07-30 (Actual); Last update posted 2021-08-23 (Actual); Status verified 2021-08

CONDITIONS: Chronic Rhinosinusitis Without Nasal Polyps (CRSsNP); Chronic Rhinosinusitis With Nasal Polyps (CRSwNP)
Keywords: GB001; Gossamer Bio; Gossamer; Nasal Polyposis; CRSwNP; CRSsNP
MeSH Terms: conditions — Nasal Polyps

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- GB001 (Experimental): GB001 40 mg once per day (QD) for 16 weeks
  Interventions: Drug: GB001
- Placebo (Placebo Comparator): Placebo QD for 16 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: GB001 — film-coated oral tablet
  Arms: GB001
Drug: Placebo — film-coated oral tablet
  Arms: Placebo

SUMMARY:
A Phase 2a, randomized, double-blind, placebo-controlled, multi-center study to evaluate the efficacy, safety, pharmacokinetics (PK), and pharmacodynamics (PD) of GB001 compared with placebo over 16 weeks of treatment in patients with chronic rhinosinusitis with or without nasal polyposis (NP).

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of chronic rhinosinusitis with nasal polyps (CRSwNP) or chronic rhinosinusitis without nasal polyps (CRSsNP) by a physician at least 12 weeks before Screening Visit
* Treated with stable intranasal corticosteroid (INCS) for at least 2 months prior to Screening Visit
* Presence of at least 2 nasal symptoms: nasal blockage/ obstruction/congestion or nasal discharge or facial pain/pressure or reduction/loss of smell
* Women of childbearing potential must use an acceptable method of contraception

Exclusion Criteria:

* Sino-Nasal Outcome Test-22 (SNOT-22) score < 20 at screening
* Asthma or chronic obstructive pulmonary disease (COPD) patients that are current smokers
* Use of other investigational drugs within 30 days, or within 5 half-lives, whichever is longer, prior to Screening Visit
* Pregnant or breastfeeding
* Pre-existing clinically important co-morbidities
* Regular use of systemic corticosteroids or immunosuppressive treatments

Other protocol-defined inclusion/exclusion criteria will apply.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 97 (Actual)
Dates: Start 2019-05-16 (Actual); Primary Completion 2020-07-09 (Actual); Study Completion 2020-08-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (38):
- United States (29):
  - Banner University of Arizona Medical Center, Tucson, Arizona
  - NEA Baptist Clinic, Jonesboro, Arkansas
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Sacramento Ear Nose and Throat Surgical and Medical Group, Inc., Roseville, California
  - Bensch Clinical Research LLC, Stockton, California
  - Yale School of Medicine, New Haven, Connecticut
  - Emory University, Atlanta, Georgia
  - Rush University Medical Center, Chicago, Illinois
  - ChicagoENT, Chicago, Illinois
  - Iowa Head & Neck, PC, Des Moines, Iowa
  - Kentuckiana Ear, Nose, and Throat, Louisville, Kentucky
  - Advanced ENT and Allergy, Louisville, Kentucky
  - Tandem Clinical Research LLC, Marrero, Louisiana
  - Chesapeake Clinical Research, Inc., White Marsh, Maryland
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Nebraska Medical Research Institute, Inc., Bellevue, Nebraska
  - BreatheAmerica Albuquerque, Albuquerque, New Mexico
  - Northwell Health at ENT and Allergy Associates, New Hyde Park, New York
  - Northwell Health at ENT and Allergy Associates, New York, New York
  - University of Rochester Medicine Otolaryngology, Rochester, New York
  - Northwell Health at ENT and Allergy Associates, White Plains, New York
  - Vital Prospects Clinical Research Institute, P.C., Tulsa, Oklahoma
  - Specialty Physician Associates, Bethlehem, Pennsylvania
  - Thomas Jefferson University Department of Otolaryngology, Philadelphia, Pennsylvania
  - Medical University of South Carolina, Department of Otolaryngology, Charleston, South Carolina
  - AARA Research Center, Dallas, Texas
  - Memorial Hermann Medical Plaza, Houston, Texas
  - Eastern Virginia Medical School, Norfolk, Virginia
  - Advanced Otolaryngology, P.C. DBA Richmond Ear, Nose and Throat, Richmond, Virginia
- Czechia (4):
  - University Hospital Hradec Kralove, Department of Otorhinolaryngology and Head and Neck Surgery, Hradec Králové
  - ENT Outpatient Clinic Pavel Navratil, Olomouc
  - Medicon a.s., Prague
  - Pulmonary Outpatient Clinic Rokycany s.r.o., Rokycany
- Ukraine (5):
  - Public Non-Profit Enterprise "Clinical Hospital of Emergency Medical Care" under Dnipro City Council, Dnipro
  - Public Non-Profit Enterprise under KRC "Regional Clinical Specialized Center for Radiation Protection of the Public", Kharkiv
  - State Institution "O.S. Kolomiychenko Institute of Otolaryngology of National Academy of Medical Sciences of Ukraine", Kyiv
  - Municipal Non-commercial Enterprise "Ternopil Municipal City Hospital #2", Ternopil
  - Public Non-Profit Enterprise "City Hospital #3" under Zaporizhia City Council, Zaporizhia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The study included a run-in period, during which eligibility for randomization was determined. 192 participants entered the run-in period, 97 of whom were randomized.
Groups:
- Placebo: Placebo once per day (QD) for 16 weeks
- GB001: GB001 40 mg QD for 16 weeks
Period: Overall Study
Arm/Group | Placebo | GB001
Started | 50 | 47
Completed | 48 | 45
Not Completed | 2 | 2
Not completed — Lost to Follow-up | 1 | 1
Not completed — Withdrawal by Subject | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | GB001 | Total
Number analyzed (Participants) | 50 | 47 | 97
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.6 (10.34) | 51.7 (11.81) | 51.7 (11.02)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 28 | 49
  Male | 29 | 19 | 48
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 47 | 41 | 88
  Black or African American | 3 | 5 | 8
  Asian | 0 | 1 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Not Hispanic or Latino | 46 | 46 | 92
  Hispanic or Latino | 4 | 1 | 5

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Week 16 in Sino-Nasal Outcome Test (SNOT) 22 Total Score
Description: The SNOT-22 is a validated questionnaire to assess the impact of chronic rhinosinusitis (CRS) on quality of life and utilizes a 2-week recall period. It is a 22-item outcome measure on a 5-point category scale applicable to sinonasal conditions and surgical treatments. The total scores range from 0 to 110 with higher total scores implying greater impact of CRS on quality of life.
Time Frame: Baseline, Week 16
Population: Intent-to-treat (ITT) population: all participants who were randomized and received at least 1 dose of study treatment. Participants with a baseline and a post-baseline value.
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Placebo | GB001
Number analyzed (Participants) | 49 | 45
score on a scale | -18.1 [-23.1 to -13.0] | -18.3 [-23.5 to -13.1]
Statistical Analysis 1: Comparison: Placebo vs GB001; Test type: Superiority; p = 0.9499, Mixed Models Analysis; Mean Difference (Net) = -0.2, 95% CI 2-sided [-7.6 to 7.1] — GB001 vs. Placebo

2. Secondary Outcome: Change From Baseline to Week 16 in Lund-Mackay Score
Description: Lund-Mackay scores are based on centralized imaging data assessments and are scored by blinded central reading at the imaging core laboratory. The Lund-Mackay system is based on localization with points given for degree of opacification: 0=normal, 1=partial opacification, 2=total opacification. These points are then applied to each sinus (maxillary, anterior ethmoid, posterior ethmoid, sphenoid, and frontal sinus) on each side. The osteomeatal complex on each side is graded as 0=not occluded, or 2=occluded. The maximum score is 12 per side, for a total score ranging from 0 to 24.
Time Frame: Baseline, Week 16
Population: ITT population: all participants who were randomized and received at least 1 dose of study treatment.
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Placebo | GB001
Number analyzed (Participants) | 50 | 47
score on a scale | -0.6 [-1.6 to 0.4] | -0.9 [-2.0 to 0.1]
Statistical Analysis 1: Comparison: Placebo vs GB001; Test type: Superiority; p = 0.6778, ANCOVA; Mean Difference (Net) = -0.3, 95% CI 2-sided [-1.8 to 1.2] — GB001 vs. Placebo

3. Secondary Outcome: Change From Baseline to Week 16 in Nasal Polyp Score (NPS)
Description: The bilateral endoscopic NPS is the sum of the right and left nostril scores, as evaluated by means of blinded, centrally read nasal endoscopy and ranges from 0 to 8. NP is graded based on polyp size: 0 = No polyps, 1 = Small polyps in the middle meatus not reaching below the inferior border of the middle turbinate, 2 = Polyps reaching below the lower border of the middle turbinate, 3 = Large polyps reaching the lower border of the inferior turbinate or polyps medial to the middle turbinate, and 4 = Large polyps causing complete obstruction of the inferior nasal cavity.
Time Frame: Baseline, Week 16
Population: ITT population: all participants who were randomized and received at least 1 dose of study treatment. Participants with nasal polyps with a baseline value.
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Placebo | GB001
Number analyzed (Participants) | 35 | 30
score on a scale | -0.8 [-1.4 to -0.3] | -0.7 [-1.3 to -0.1]
Statistical Analysis 1: Comparison: Placebo vs GB001; Test type: Superiority; p = 0.7914, Mixed Models Analysis; Mean Difference (Net) = 0.1, 95% CI 2-sided [-0.7 to 0.9] — GB001 vs. Placebo

4. Secondary Outcome: Time to First Response in NPS
Description: Response was defined as ≥ 1-point improvement from baseline.
  The bilateral endoscopic NPS is the sum of the right and left nostril scores, as evaluated by means of blinded, centrally read nasal endoscopy and ranges from 0-8. NP is graded based on polyp size: 0 = No polyps, 1 = Small polyps in the middle meatus not reaching below the inferior border of the middle turbinate, 2 = Polyps reaching below the lower border of the middle turbinate, 3 = Large polyps reaching the lower border of the inferior turbinate or polyps medial to the middle turbinate, and 4 = Large polyps causing complete obstruction of the inferior nasal cavity.
Time Frame: up to Week 16
Population: ITT population: all participants who were randomized and received at least 1 dose of study treatment. Participants with nasal polyps.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Placebo | GB001
Number analyzed (Participants) | 35 | 32
weeks | 16.43 [8.571 to NA] — NA (Not Available) indicates the value is not estimable due to an insufficient number of observed events. | 16.14 [8.143 to NA] — NA (Not Available) indicates the value is not estimable due to an insufficient number of observed events.
Statistical Analysis 1: Comparison: Placebo vs GB001; Test type: Superiority; p = 0.8916, Regression, Cox; Hazard Ratio (HR) = 0.944, 95% CI 2-sided [0.410 to 2.173] — GB001 vs Placebo

5. Secondary Outcome: Change From Baseline to Week 16 in Morning (AM) Nasal Congestion (NC) Score
Description: AM NC score was assessed using a 0 to 3 categorical scale (where 0 = no symptoms, 1 = mild symptoms, 2 = moderate symptoms and 3 = severe symptoms).
Time Frame: Baseline, Week 16
Population: ITT population: all participants who were randomized and received at least 1 dose of study treatment. Participants with a baseline value.
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Placebo | GB001
Number analyzed (Participants) | 50 | 46
score on a scale | -0.733 [-0.917 to -0.549] | -0.543 [-0.738 to -0.347]
Statistical Analysis 1: Comparison: Placebo vs GB001; Test type: Superiority; p = 0.1635, Mixed Models Analysis; Mean Difference (Net) = 0.191, 95% CI 2-sided [-0.077 to 0.459] — GB001 vs. Placebo

6. Secondary Outcome: Change From Baseline to Week 16 in AM Total Symptom Score (TSS)
Description: AM TSS is the sum of the scores from the 4 AM symptom categories (congestion and/or obstruction, anterior rhinorrhea, posterior rhinorrhea, loss of sense of smell) and ranges from 0-12. Each symptom category was assessed using a 0 to 3 categorical scale (where 0 = no symptoms, 1 = mild symptoms, 2 = moderate symptoms and 3 = severe symptoms).
Time Frame: Baseline, Week 16
Population: as for outcome 5
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Placebo | GB001
Number analyzed (Participants) | 50 | 46
score on a scale | -2.499 [-3.130 to -1.869] | -1.867 [-2.526 to -1.209]
Statistical Analysis 1: Comparison: Placebo vs GB001; Test type: Superiority; p = 0.1742, Mixed Models Analysis; Mean Difference (Net) = 0.632, 95% CI 2-sided [-0.280 to 1.544] — GB001 vs. Placebo

7. Secondary Outcome: Change From Baseline to Week 16 in University of Pennsylvania Smell Identification Test (UPSIT) Score
Description: The UPSIT test consists of four booklets, each containing 10 odorants with one odorant per page. The test-time is about 15 minutes. The stimuli are embedded in 10-50 μm diameter plastic microcapsules on brown strips at the bottom of each page. Above each odorant strip is a multiple-choice question with four alternative words to describe the odor. The participant is asked to release the odorant by rubbing the brown-strip with the tip of a pencil and to indicate which of 4 words best describes the odor. An UPSIT result is scored from 0 to 40 where a higher score indicates better olfaction.
Time Frame: Baseline, Week 16
Population: as for outcome 5
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Placebo | GB001
Number analyzed (Participants) | 49 | 47
score on a scale | 1.5 [-0.3 to 3.2] | 2.3 [0.5 to 4.2]
Statistical Analysis 1: Comparison: Placebo vs GB001; Test type: Superiority; p = 0.4851, ANCOVA; Mean Difference (Net) = 0.9, 95% CI 2-sided [-1.6 to 3.4] — GB001 vs. Placebo

8. Secondary Outcome: Time to First Chronic Rhinosinusitis (CRS) Exacerbation
Description: Chronic rhinosinusitis exacerbation is defined as deterioration of CRS symptoms requiring treatment with an antibiotic, an anti-inflammatory drug, or a symptom reliever; an Emergency Department visit; or hospitalization.
Time Frame: up to Week 16
Population: ITT population: all participants who were randomized and received at least 1 dose of study treatment.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Placebo | GB001
Number analyzed (Participants) | 50 | 47
weeks | NA [NA to NA] — NA (Not Available) indicates the value is not estimable due to an insufficient number of observed events. | NA [NA to NA] — NA (Not Available) indicates the value is not estimable due to an insufficient number of observed events.
Statistical Analysis 1: Comparison: Placebo vs GB001; Test type: Superiority; p = 0.3898, Regression, Cox; Hazard Ratio (HR) = 0.544, 95% CI 2-sided [0.136 to 2.178] — GB001 vs Placebo

9. Secondary Outcome: Percentage of Participants With a Treatment-Emergent Adverse Event (AE)
Description: An adverse event (AE) is any untoward medical occurrence in a participant, whether or not considered related to study drug. Abnormal laboratory test results or other safety assessments, including those that worsened from baseline, that were considered clinically significant in the medical and scientific judgment of the investigator were to be reported as AEs.
Time Frame: From first dose of study drug through Week 20
Population: Safety Population: all participants who received at least 1 dose of study treatment.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | GB001
Number analyzed (Participants) | 50 | 47
percentage of participants | 36.0 | 44.7

ADVERSE EVENTS:
Time Frame: From first dose of study drug through Week 20
Arm/Group | Placebo | GB001
All-Cause Mortality (participants affected / at risk) | 0/50 | 0/47
Serious Adverse Events (participants affected / at risk) | 0/50 | 1/47
Other Adverse Events (participants affected / at risk) | 10/50 | 12/47
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=50) | GB001 (N=47)
Endometriosis (Reproductive system and breast disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=50) | GB001 (N=47)
Nasopharyngitis (Infections and infestations) | 3 | 2
Headache (Nervous system disorders) | 3 | 5
Asthma (Respiratory, thoracic and mediastinal disorders) | 2 | 3
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2020-04-16): https://cdn.clinicaltrials.gov/large-docs/62/NCT03956862/Prot_000.pdf
  • Statistical Analysis Plan (2020-09-01): https://cdn.clinicaltrials.gov/large-docs/62/NCT03956862/SAP_001.pdf